CLINICAL TRIAL: NCT04691882
Title: Factors That Determine the Responses to Meal Ingestion: Effect of Abdominal Wall Activity
Brief Title: Effect of Abdominal Wall Activity on the Responses to Meal Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PR(AG)338/2016K
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: meal ingestion; postprandial responses; hedonic sensations; homeostatic sensations; abdominal wall activity; abdominal distension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic contraction (Experimental)
  Interventions: Behavioral: Diaphragmatic contraction
- Diaphragmatic relaxation (Active Comparator)
  Interventions: Behavioral: Diaphagmatic relaxation

INTERVENTIONS:
Behavioral: Diaphragmatic contraction — Sequential periods (30 s) of voluntary diaphragmatic contraction after meal ingestion
  Arms: Diaphragmatic contraction
Behavioral: Diaphagmatic relaxation — Sequential periods (30 s) of voluntary diaphragmatic relaxation after meal ingestion
  Arms: Diaphragmatic relaxation

SUMMARY:
Meal ingestion induces sensations that are influenced by a series of conditioning factors. Aim: to determine the effect of abdominal wall activity on the responses to a standard probe meal. Study in healthy subjects comparing postprandial digestive sensations (abdominal bloating and digestive well-being) during consecutive maneuvers of diaphragmatic contraction (i.e. descent) versus diaphragmatic relaxation (i.e. ascent) in a cross-over randomized design. Primary outcome: effect of somatic maneuvers on abdominal bloating sensation; secondary aim: effect on digestive well-being.

Participants (16 women) will be instructed to eat a standard dinner the day before, to consume a standard breakfast at home after overnight fast, and to report to the laboratory, where the test meal will be administered 4 h after breakfast. Studies will be conducted in a quiet, isolated room. Participants will be taught to produce diaphragmatic contraction and visible abdominal distention. A probe meal up to maximal satiation will be administered to induce abdominal fullness/bloating sensation; immediately after ingestion, bloating sensation (from 0 to 10) and digestive well-being (from -5 to +5) will be scored during 8 alternating episodes (30 s each) in random sequence of diaphragmatic contraction (abdominal distension) versus diaphragmatic relaxation.

ELIGIBILITY:
Inclusion Criteria:

* non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Changes in abdominal fullness/bloating sensation induced by the probe meal | 10 min
  Effect of abdominal wall activity on abdominal fullness/bloating [measured by 10 cm scale graded from 0 (not at all) to 10 (very much)]

SECONDARY OUTCOMES:
Changes in digestive well-being sensation induced by the probe meal | 10 min
  Effect of abdominal wall activity on digestive well-being [measured by 10 cm scale graded from -5 (extremely unpleasant sensation) to +5 (extremely unpleasant extremely pleasant sensation)]

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Livovsky DM, Pribic T, Azpiroz F. Food, Eating, and the Gastrointestinal Tract. Nutrients. 2020 Apr 2;12(4):986. doi: 10.3390/nu12040986. PMID 32252402
- [Derived] Livovsky DM, Barber C, Barba E, Accarino A, Azpiroz F. Abdominothoracic Postural Tone Influences the Sensations Induced by Meal Ingestion. Nutrients. 2021 Feb 18;13(2):658. doi: 10.3390/nu13020658. PMID 33670508